CLINICAL TRIAL: NCT00549289
Title: Study of Cyclosporine in the Treatment of Dry Eye Syndrome (ST-603-006)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sirion Therapeutics, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: ST-603-006
Record Dates: First submitted 2007-10-24; First posted 2007-10-25 (Estimated); Last update posted 2007-10-25 (Estimated); Status verified 2007-10

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporine

INTERVENTIONS:
Drug: cyclosporine A

SUMMARY:
The purpose of this phase III, open-label study is to determine the safety and tolerability of cyclosporine in the treatment of dry eye syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of dry eye syndrome

Exclusion Criteria:

* Intraocular or refractive surgery in the study eye within 3 months prior to study start
* Unwilling to discontinue use of contact lenses during the study
* Pregnancy or lactation

Min Age: 2 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Roger Vogel, Study Chair — Sirion Therapeutics
Locations (1):
- Clayton Eye Center, Morrow, Georgia, United States